CLINICAL TRIAL: NCT03452514
Title: Prospective Longitudinal Blinded Observational Diagnostic Study - Addition of microRNA Blood Test to Lung Cancer Screening Low Dose CT
Brief Title: Addition of microRNA Blood Test to Lung Cancer Screening Low Dose CT
Status: Completed | Type: Observational
Sponsor: Hummingbird Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: HMBDx USA-0001
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be drawn from all patients at the time of study enrollment prior to LDCT scanning (10cc blood divided into 2 PAXgene tubes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Low Dose CT (LDCT) Scan: Individuals undergoing their first or subsequent annual LDCT screening study
- Cohort 2 - Diagnostic CT Scan: Individuals referred for a follow-up diagnostic chest CT scan due to a lung-RADS category 3 or 4 result on a previous LDCT scan

SUMMARY:
To demonstrate that the specificity of the Hummingbird microRNA profile for the diagnosis of lung cancer in a cohort of patients who meet current eligibility criteria for lung cancer screening in the U.S. is superior to the specificity of LDCT.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, blinded, observational diagnostic study on 400 individuals undergoing lung cancer screening with low-dose computed tomography (LDCT).

There will be two patient cohorts: Cohort 1: individuals undergoing their first or subsequent annual LDCT screening study; and Cohort 2: individuals referred for a follow-up diagnostic chest CT scan due to a lung-RADS category 3 or 4 result on a previous LDCT scan.

At study enrollment a blood sample will be drawn prior to the LDCT scan. On this blood sample a novel lung cancer test relying on microRNA signatures will be evaluated. The results will be compared with the CT scan results and follow-up tests including pathology. Histologic results and follow-up data will be collected on all patients for a minimum of 12 months post-enrollment. During the follow-up period, the results of all diagnostic chest CT scans, lung biopsies or lung resections will be captured from the Partners electronic medical record and entered into the case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing LDCT screening for lung cancer.
2. Subject is 55 to 80 years of age.
3. Subject has a minimum 30 pack-year smoking history.
4. Subject has not quit smoking more than 15 years ago.
5. Subject is without symptoms attributable to lung cancer.
6. Subject is able and willing to provide informed consent.

Exclusion Criteria:

1. Subject has a history of lung, gastrointestinal, hematological, breast, thyroid, or genitourinary cancers within the past ten years.
2. Subject is known to be infected with HIV, HBV, HCV, or tuberculosis or any other Biosafety Level 3 (BSL III) pathogen infections.

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible for Lung Cancer Screening as per the National Lung Screening Trial (NLST) Guidelines
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Specificity of HMBDx microRNA Test for Lung Cancer | 12 months
  The reference standard will be the combination of all available diagnostic information (LDCT, subsequent diagnostic imaging studies, biopsy results and surgical pathology results) obtained during at least 12 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Amita Sharma, MD, Study Director — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zyla J, Dziadziuszko R, Marczyk M, Sitkiewicz M, Szczepanowska M, Bottoni E, Veronesi G, Rzyman W, Polanska J, Widlak P. miR-122 and miR-21 are Stable Components of miRNA Signatures of Early Lung Cancer after Validation in Three Independent Cohorts. J Mol Diagn. 2024 Jan;26(1):37-48. doi: 10.1016/j.jmoldx.2023.09.010. Epub 2023 Oct 20. PMID 37865291